CLINICAL TRIAL: NCT00809718
Title: The Effect of Rifapentine on Plasma Concentrations of Raltegravir
Brief Title: The Effect of Rifapentine on Raltegravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Centers for Disease Control and Prevention (U.S. Federal Agency); VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TBTC 29RR
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: Raltegravir; Pharmacokinetics; Rifapentine; Drug Kinetics
MeSH Terms: interventions — Raltegravir Potassium; rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- raltegravir and rifapentine (Other): Concomitant administration of raltegravir and rifapentine in healthy volunteers
  Interventions: Drug: Raltegravir and rifapentine

INTERVENTIONS:
Drug: Raltegravir and rifapentine — Period 1- Raltegravir 400 mg q12h by mouth for 4 days
  Period 2- Rifapentine 900 mg taken by mouth once per week for 3 doses and raltegravir 400 mg q12h by mouth for 4 days
  Period 3- Rifapentine 600 mg taken by mouth once daily for 5 of 7 days per week for 10 doses and raltegravir 400 mg q12h by mouth for 4 days
  Other Names: Isentress - Raltegravir; Priftin - Rifapentine

SUMMARY:
The aim of this study is to study the effect of rifapentine on plasma concentrations of raltegravir.

DETAILED DESCRIPTION:
Primary Objective

To compare the pharmacokinetics parameter values (geometric mean Cmin and AUC) of raltegravir at 400 mg q12h alone to raltegravir at 400 mg q12h co-administered in combination with rifapentine 900 mg once weekly, and to raltegravir at 400 mg q12h co-administered in combination with rifapentine 600 mg per day, 5 days per week.

Secondary Objective

To assess the tolerability and safety of concomitant administration of raltegravir and rifapentine in healthy volunteers.

Design

This study is a three-period, one-sequence, open label, pharmacokinetic study of the raltegravir-rifapentine interactions in healthy, male and female volunteers. Up to 21 subjects may be enrolled to achieve the estimated sample size of 16 completing subjects. All study medication will be self-administered except on the days of pharmacokinetic sampling. All subjects will participate in three sampling periods and be studied in a day clinic or be admitted overnight to a hospital.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female age > 18 years in good health
* Provision of informed consent for the study.
* HIV-uninfected. A prior negative HIV test (ELISA) must be obtained before enrollment.
* Willingness to have PK sampling in a day clinic or to be admitted overnight to a hospital on three occasions.
* Women of child-bearing potential must agree to practice an adequate method of birth control during the study and for 30 days after the last dose of study medication. Barrier methods of contraception or abstinence from sexual activity are satisfactory methods of birth control.
* Karnofsky score ≥ 90.
* Laboratory screening before enrollment:

  * Hematocrit > 30 percent (most recent value)
  * AST < 2 times the upper limit of normal
  * ALT < 2 times the upper limit of normal
  * Bilirubin < 2 times the upper limit of normal
  * Creatinine < 1.5 times the upper limit of normal
  * Negative urine drug screen

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Use of a medication or food that has the potential to alter the concentrations of raltegravir or rifapentine, within the 14 days prior to or during the periods of pharmacokinetic monitoring.
* Known intolerance to raltegravir or rifamycin antibiotics or prior use in the last 30 days.
* Weight less than 46 kg or greater than 102 kg.
* Prior gastrointestinal surgery.
* Infection with Hepatitis B or Hepatitis C by serologies.
* Co-morbidity for which concomitant, current medications are taken regularly. If concomitant medications are taken intermittently, these medications should not have potential to alter the concentrations of raltegravir or rifapentine.
* Current imprisonment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Raltegravir pharmacokinetics (Cmin and AUC) | Eight weeks

SECONDARY OUTCOMES:
Tolerability and safety of concomitant raltegravir and rifapentine administration | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc Weiner, M.D., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Audie L Murphy Veterans Administration Hospital, San Antonio, Texas
  - University of Texas Health Science Center, San Antonio, Texas

REFERENCES:
- [Derived] Weiner M, Egelund EF, Engle M, Kiser M, Prihoda TJ, Gelfond JA, Mac Kenzie W, Peloquin CA. Pharmacokinetic interaction of rifapentine and raltegravir in healthy volunteers. J Antimicrob Chemother. 2014 Apr;69(4):1079-85. doi: 10.1093/jac/dkt483. Epub 2013 Dec 15. PMID 24343893